CLINICAL TRIAL: NCT06023966
Title: A Clinical Prospective Study to Validate a Risk Scoring Model for the Hepatic Metastases From Gastric Cancer After Curative Surgery
Brief Title: A Clinical Prospective Study to Validate a Risk Scoring Model for the HMGC After Curative Surgery
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DJY003
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2023-08

CONDITIONS: Predictive Cancer Model; Hepatic Metastasis; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with HMGC: patients with gastric cancer who developed hepatic metastasis after curative gastrectomy
- without HMGC: patients with gastric cancer who did not developed hepatic metastasis after curative gastrectomy

SUMMARY:
A previous study of investigators established a risk scoring model for occurrence of postoperative hepatic metastases in patients who underwent curative gastrectomy directly without neoadjuvant therapy. In order to further validate the clinical applicability of abovementioned model, investigators designed this prospective study, which also included patients who received neoadjuvant therapy before surgery, with the aim of exploring the applicability of the risk scoring model to this group of patients.

DETAILED DESCRIPTION:
The study was a single-centre, prospective study. Prospectively collected data were used to analyze the consistency between the actual outcomes of patients with or without hepatic metastases after curative gastrectomy and the predicted outcomes of the risk scoring model, in order to assess the clinical applicability of the model. In addition, analyses were performed to compare the differences in the risk of hepatic metastasis and the time interval of occurrence between patients who did not receive neoadjuvant therapy and those who received neoadjuvant therapy, as well as between patients with different outcomes after receiving neoadjuvant therapy (TRG 0-1 vs. TRG 2-3 in postoperative pathology).

ELIGIBILITY:
Inclusion Criteria:

1. Received curative gastrectomy (D2 lymph node dissection);
2. Gastric cancer without distant organ metastasis, distant lymph node metastasis and peritoneal implantation (M0) confirmed by postoperative pathology;
3. No hepatic tumors and other occupying diseases, no chronic diseases such as cirrhosis and hepatitis, no hepatic schistosomiasis, no hepatic echinococcosis, no hepatic tuberculosis, and no severe fatty liver disease before the curative surgery;
4. No history of intraperitoneal chemotherapy;
5. No other serious concomitant diseases with satisfactory organ function;
6. No history of other malignant tumors;
7. Comply with the protocol during the whole study period;
8. Sign informed consent and permission of withdraw in the whole study period;
9. Estimation the overall survival after surgery no less than 12 months;
10. Consent to analysis of clinicopathological data and prognostic follow up;
11. Karnofsky Performance Scores (KPS) more than 60.

Exclusion Criteria:

1. Special histological types of gastric cancer (neuroendocrine, squamous, squamous cell, hepatoid adenocarcinoma or others);
2. Gastro-esophageal junction cancer;
3. Severe congestive heart failure, frequent arrhythmia, or myocardial infarction within 12 months;
4. Immunosuppressive therapists for organ transplantation;
5. Seriously uncontrolled recurrent infection;
6. History of other malignancies;
7. No abilities of self-knowledge or mental disorders;
8. Combination of other serious diseases;
9. Concurrent participation in other clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patietns who were diagnosed with gastric cancer pathologically and underwent curative gastrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
hepatic metastasis | 2 years after curative surgery
  Postoperative telephone follow-up was performed in patients with gastric cancer undergoing curative gastrectomy to determine the occurrence of hepatic metastasis.

SECONDARY OUTCOMES:
interval between the surgery and hepatic metastasis | 2 years after curative surgery
  Postoperative telephone follow-up was performed in patients with gastric cancer undergoing curative gastrectomy to determine the interval between the gastrectomy and development of hepatic metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2023-04-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT06023966/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT06023966/SAP_001.pdf
  • Informed Consent Form (2023-04-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT06023966/ICF_002.pdf